CLINICAL TRIAL: NCT00340990
Title: Pilot Study of CD4+ T Cell Immune Responses to Mycobacterium Tuberculosis
Brief Title: Immune Responses to Mycobacterium Tuberculosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904009; 04-I-N009
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2015-11-27

CONDITIONS: Mycobacterium Tuberculosis
Keywords: Tuberculosis; HIV; CD4+ T Cell; Interferon-Gamma; Lymphocyte Proliferation
MeSH Terms: conditions — Tuberculosis

SUMMARY:
This study, conducted at the University of Mali in the capital city of Bamako, will investigate how the body reacts to infection with Mycobacterium tuberculosis (MTB), the organism that causes tuberculosis. Tuberculosis is a major global health problem whose solution requires development of an effective vaccine. However, incomplete understanding of how immunity to MTB is acquired and measured limits vaccine development. This study will focus on certain immune system cells - CD4+ T cells - that appear to be very important in fighting tuberculosis.

Individuals 16 years of age and older who have or have not been exposed to either tuberculosis or HIV, or both, may be eligible for this study. Candidates will be screened with a medical history, physical examination, blood tests, review of medical records and laboratory tests, and, if medically indicated, a chest x-ray. Individuals whose medical records indicate a past history of tuberculosis or a positive test for exposure to tuberculosis will have a tuberculin skin test. For this test, a few drops of fluid are placed under the skin to see if the immune system reacts to the substance, indicating previous exposure to MTB.

Participants will come to the University of Mali 10 times over a 1-year period - 7 times within the first 3 months of the study and then once every 3 months until 1 year after enrollment. At each study visit, they will be asked about their medical history and will donate 75 milliliters (about 1/3 cup) of blood, totaling 830 mL over the entire year. More blood may be requested if the participant's immune system reacts strongly to MTB in laboratory tests. No more than 450 mL (2 cups) of blood would be collected every 6 weeks; this amount is the Red Cross limit for regular blood donations every 6 weeks.

The blood samples will be used for tests that measure the level of immunity to tuberculosis. Genetic tests may be performed on blood cells to help interpret special tests of immunity. Because HIV-infected people are included in the study, the findings may also provide information on how HIV renders vulnerability to opportunistic infections, including tuberculosis.

DETAILED DESCRIPTION:
Tuberculosis is a daunting global health problem. The solution requires development of an effective vaccine. But incomplete understanding of Mycobacterium tuberculosis (MTB) immunity-how it is acquired, how it is measured-limits vaccine development to empiric rather than rational approaches. New perspectives are needed. Most individuals infected with MTB never actually develop active tuberculosis. Similarly, most individuals with treated tuberculosis or BCG vaccination are also protected from subsequent disease. These individuals may be said to be immune. One approach to obtaining greater understanding of MTB immunity is to study these individuals to discover mechanisms of immunity that mediate their protection from disease. Because it is already known that CD4+ T cells are a critical component of MTB immunity, studying CD4+ T cell responses to MTB infection in immune individuals is a reasonable starting point. To determine which CD4+ T cell subsets and which CD4+ T cell immune responses are important, we will compare individuals with prior exposure (immunity) to MTB to individuals with active tuberculosis. Because HIV infection interferes with the CD4+ T cell response to MTB, it dramatically increases the risks for acquiring MTB infection and for developing disease. Under these circumstances it is easier to discern mechanisms relevant to MTB immunity because of exaggerated MTB-specific responses. In this study we aim to identify CD4+ T cell subsets and responses that correlate with MTB immunity. We anticipate that these correlations will yield new insight into mechanisms of MTB immunity that will be relevant to vaccine development. In addition, by examining MTB immunity in the setting of HIV coinfection, we anticipate new insights into mechanisms of how HIV causes disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ability to sign informed consent and willingness to comply with study requirements (including storage of blood specimens for future research on HIV, AIDS, MTB or the immune system).

CATEGORY-SPECIFIC MTB INCLUSION CRITERIA:

Group A (HIV-/MTB[BCG]) HIV ELISA(2) negative; BCG vaccinated with TST(2) less than 15 mm

Group B (HIV+/MTB[BCG]) HIV ELISA/WB(2) positive; BCG vaccinated with TST less than 5 mm

Group C (HIV-/MTB[pulm]) HIV ELISA negative; pulmonary MTB

Group D (HIV-/MTB[diss]) HIV ELISA negative; disseminated MTB

Group E (HIV+/MTB[pulm]) HIV ELISA/WB positive; pulmonary MTB

Group F (HIV+/MTB[diss]) HIV ELISA/WB positive; disseminated MTB

EXCLUSION CRITERIA:

Age less than 18 years (because of the risk for inducing protocol-related anemia)

Hg less than 7.5 g/dL

Latent MTB infection (as evidenced by a TST greater than 5 mm if HIV infected or greater than 15 mm if HIV uninfected) for arms A and B only.

Past history of treated MTB infection

Known or underlying bleeding disorder (due to risk of bleeding from venipuncture)

Psychiatric illness that might interfere with study compliance

Use of immunomodulators (including corticosteroids and IL-2) or cytotoxic agents (including hydroxyurea) within 45 days of signing consent and at any time during study

Small or difficult to access antecubital veins that make venipuncture difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2003-10-06; Study Completion 2015-11-27

CONTACTS AND LOCATIONS:
Overall Officials: Sophia B Siddiqui, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Mali, Bamako, Mali

REFERENCES:
- [Background] Ellner JJ. Review: the immune response in human tuberculosis--implications for tuberculosis control. J Infect Dis. 1997 Nov;176(5):1351-9. doi: 10.1086/514132. No abstract available. PMID 9359738
- [Background] Orme IM, Andersen P, Boom WH. T cell response to Mycobacterium tuberculosis. J Infect Dis. 1993 Jun;167(6):1481-97. doi: 10.1093/infdis/167.6.1481. PMID 8501346
- [Background] Sallusto F, Lenig D, Forster R, Lipp M, Lanzavecchia A. Two subsets of memory T lymphocytes with distinct homing potentials and effector functions. Nature. 1999 Oct 14;401(6754):708-12. doi: 10.1038/44385. PMID 10537110